CLINICAL TRIAL: NCT03292757
Title: FLuOrescence to Identify the Thoracic Duct During Oesophageal Resections
Brief Title: FLOTOR Pilot Study
Acronym: FLOTOR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Thomas Barnes, Clinical Research Fellow, Oxford University Hospitals NHS Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12968
Record Dates: First submitted 2017-09-18; First posted 2017-09-26 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Chylothorax; Esophageal Cancer; Thoracic Duct Intra-Operative Injury
Keywords: Fluorescence
MeSH Terms: conditions — Chylothorax; Esophageal Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenteric ICG (Experimental): Indocyanine green injected into the small bowel mesentery during oesophagectomy.
  Interventions: Drug: Indocyanine Green
- Feeding jejunostomy ICG (cream) (Experimental): Indocyanine green mixed with cream infiltrated into the feeding jejunostomy.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Fluorescent dye - indocyanine green
  Other Names: ICG

SUMMARY:
This is a non-randomised study assessing the technique of using indocyanine green as a fluorescent dye to highlight the thoracic duct during oesophectomy.

DETAILED DESCRIPTION:
The thoracic duct is the largest vessel of the lymphatic system in the body. It transports chyle (a liquid containing both lymph and emulsified fats) from most of the body, including the gastrointestinal tract, into the left internal jugular vein. It is largely located in the thorax and is at risk of injury during the thoracic part of an oesophagectomy.

The reported incidence of thoracic duct injury during oesophagectomy is between 0.2 and 10.5%, although it may be under-reported in the literature. A review of prospective collected complication data from 292 consecutive oesophagectomies performed in Oxford over a 5 year period revealed a chyle leak rate of 9.9%. Chyle leak was associated in a doubling of median length of post-operative stay from 8 to 16 days in these patients. Chylothorax has been associated with a mortality of up to 30%.

Over the years, a number of attempts have been made to visualise chyle leakage following thoracic duct injury including administration of enteral fat containing feed (e.g. double cream), methylene blue and lymphoscintigraphy, but no studies have been published showing a mechanism to aid thoracic duct identification at the index operation, and so prevent injuries.

Fluorescence is a technique which uses fluorescent dyes (fluorophores) that emit invisible (near infra-red (NIR)) light when they are excited by light at a particular wavelength. In order to use this technique, a fluorescence-enabled camera is required in order to shine light at that particular wavelength on the fluorophore and to capture the light emitted. This is then displayed on a screen for the surgeon to see.

Indocyanine green (ICG) is a fluorescent molecule that is approved by the FDA (Food and Drug Administration) and the MHRA for use in humans. It is a widely used near infra-red dye for numerous operations. Near infra-red guided lymphatic mapping with ICG has gained much attention over recent years and its use has widely been published in breast and colorectal surgery. ICG has also been successfully used to identify the thoracic duct in a number of case reports in both adults and children.

ICG can be injected into the small bowel mesentery to aid identification of thoracic duct injury at re-exploration. This study aims to assess the feasibility of using ICG fluorescence to identify the thoracic duct during oesophagectomy, with the eventual aim of developing its routine use to prevent thoracic duct injuries.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Undergoing elective oesophagectomy

Exclusion Criteria:

* Known allergy to iodine or ICG
* Female patient who is pregnant, planning pregnancy or breastfeeding
* Patient has a lactose intolerance (excluded only from receiving cream method)
* Known significant liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Number of thoracic ducts seen under fluorescence versus number of thoracic ducts seen with white light. (Change over time) | 0, 5, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 120, 180, 240 minutes post dose
  Thoracic duct visualised fluorescence assessment

SECONDARY OUTCOMES:
Signal to background ratio of fluorescence in thoracic ducts between 2 methods of ICG administration. | 0, 5, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 120, 180, 240 minutes post dose
  Thoracic duct fluorescence levels between methods of ICG administration
Signal to background ratio of fluorescence in thoracic ducts between dosing levels. | 0, 5, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 120, 180, 240 minutes post dose
  Thoracic duct fluorescence levels between ICG doses

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gillies, MBChB, Principal Investigator — Consultant Upper GI Surgeon; Thomas Barnes, MBChB, Principal Investigator — Clinical Research Fellow
Locations (1):
- Department of Upper GI Surgery, Oxford University Hospitals, Headington, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data

REFERENCES:
- [Derived] Barnes TG, MacGregor T, Sgromo B, Maynard ND, Gillies RS. Near infra-red fluorescence identification of the thoracic duct to prevent chyle leaks during oesophagectomy. Surg Endosc. 2022 Jul;36(7):5319-5325. doi: 10.1007/s00464-021-08912-1. Epub 2021 Dec 14. PMID 34905086